CLINICAL TRIAL: NCT02524691
Title: Efficacy Study of Rapid Immunoassay Diagnostic Test Utilizing PP12 and AFP, ROM Plus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinical Innovations, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-002-RP
Record Dates: First submitted 2015-07-31; First posted 2015-08-17 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: PROM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Use of Rapid Immunoassay Tests for the Detection of PROM — Patient will undergo both rapid immunoassay tests for the detection of PROM and the standard of care for the diagnosis of PROM using a sterile speculum (SSE). Women who cannot be confirmed clinically by the SSE will undergo an ultrasound evaluation to determine the amniotic fluid index. The patient will be treated according to the results of the SSE and ultrasound, not the results of rapid immunoassay tests. The provider conducting the SSE will be blinded to the results of the rapid immunoassay tests.
  Other Names: ROM Plus; Amnisure

SUMMARY:
The study is designed to establish the level of agreement between the ROM Plus test and the diagnosis of ROM as defined by the patient's clinical course, with respect to a population of pregnant women who present to the clinical site with signs and symptoms suggestive of ROM.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM), defined as spontaneous rupture of membranes (ROM) before the onset of uterine contractions, is one of the most common diagnostic dilemmas in contemporary obstetrical practice. Premature rupture of membranes can occur at any gestational age, and preterm PROM (PPROM, defined as PROM before 37 weeks) is responsible for 20-40% of preterm births. Early and accurate diagnosis of PROM would allow for gestational age-specific obstetrical interventions designed to optimize perinatal outcome and minimize serious complications such as cord prolapse, preterm delivery, fetal distress and infectious morbidity (chorioamnionitis, neonatal sepsis). Conversely, a false-positive diagnosis of PROM may lead to unnecessary obstetric interventions, including hospitalization, administration of antibiotics and corticosteroids, and even induction of labor. Therefore, the correct and timely diagnosis of this disorder is of critical importance to the clinician because PROM and PPROM may be associated with serious maternal and neonatal consequences.

The diagnosis of fetal membrane rupture is conventionally made using a clinical assessment. The most common method of diagnosis includes the sterile speculum exam (SSE) which includes visual inspection of pooling of fluid in the posterior fornix, a nitrazine/pH testing of the vaginal environment, and a microscopic evaluation of the collected specimen (ferning). If during the sterile speculum exam, the clinician observes amniotic fluid leaking from the cervical os, then the diagnosis of rupture can be made without the three additional evaluations. Although the SSE approach is considered an acceptable standard, it requires an intrusive (speculum) examination and may not provide a rapid or accurate diagnosis.

The literature has shown the SSE to have limitations in terms of diagnostic accuracy, cost and technical ease. The test becomes progressively less accurate when more than one hour has elapsed after the membranes are ruptured. The nitrazine assessment, which is the most common method of determining the status of the membranes in hospitals today, has a sensitivity reported between 90-97%, but a specificity as low as 16-70%. The poor specificity is thought to be due to a high rate of false-positives caused by cervicitis, vaginitis, and contamination with blood, urine, semen and antiseptic agents. The reported sensitivity and specificity for the fern test are also less than adequate, at 51% and 70% respectively.

As a result, rapid, point of care, qualitative immunochromatographic tests (ie., ROM Plus®, Amnisure®) have recently gained popularity as aids in the diagnosis of fetal membrane rupture. These tests are designed to detect proteins found in amniotic fluid at high concentrations. One such test, ROM Plus, uses a unique monoclonal/polyclonal antibody approach to detect two different proteins found in amniotic fluid at high concentrations. ROM Plus detects Placental Protein-12 (PP-12, also known as Insulin-like Growth Factor Binding Protein-1) as well as Alpha Fetoprotein (AFP). The combination of PP12 and AFP were chosen not only because of their robust historical literature support as ideal protein markers for amniotic fluid, but also their unique characteristics. PP12 is synthesized by the decidua of the placenta and reaches a very high concentration level in the amniotic fluid early in the first trimester and stays at that level until delivery. AFP is synthesized by the fetal liver and yolk sac and reaches its peak concentration late in the second trimester/early third trimester. This increases the chance that the proteins will be detected, especially in the preterm patients, when the diagnosis of ROM is most crucial. Amnisure uses a monoclonal/monoclonal antibody approach to detect one protein, Placenta-Alpha Microglobulin-1 (PAMG-1).

This study is designed to assess the performance (sensitivity, specificity, PPV, NPV) of ROM Plus and Amnisure as compared to the standard clinical assessment including but not limited to nitrazine, ferning and/or sterile speculum exam confirmed by a thorough chart review after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >15 weeks gestation undergoing an evaluation for suspected ROM, as indicated by standard site procedures (multiple gestations will not be excluded).
* Patients (or their legal representatives) who are willing to voluntarily agree to sign a consent form.

Exclusion Criteria:

* Known placental previa
* Active vaginal bleeding (≥ menstrual period)
* Individuals < 18 years of age.
* Patients (or their legal representatives) who are unwilling to voluntarily agree to sign a consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women undergoing an evaluation for suspected ROM.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The level of agreement between the ROM Plus test and the diagnosis of ROM as defined by the patient's clinical course, with respect to a population of pregnant women who present to the clinical site with signs and symptoms suggestive of ROM | 3 months

SECONDARY OUTCOMES:
Number of tests results from the ROM Plus test that provide the same result as the Amnisure test | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross W McQuivey, MD, Study Chair — Clinical Innovations, LLC
Locations (3):
- United States (3):
  - Christiana Care Health Services, Newark, Delaware
  - Cooper Health System, Camden, New Jersey
  - Intermountain Healthcare, Salt Lake City, Utah